CLINICAL TRIAL: NCT01638533
Title: A Phase 1 and Pharmacokinetic Single Agent Study of Romidepsin in Patients With, Lymphomas, Chronic Lymphocytic Leukemia, and Select Solid Tumors and Varying Degrees of Liver Dysfunction
Brief Title: Romidepsin in Treating Patients With Lymphoma, Chronic Lymphocytic Leukemia, or Solid Tumors With Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01040; NCI-2012-01040 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737061; NCI-2013-01545; J11105; NA_00052587; 9008 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9008 (Other: CTEP); U01CA132123 (NIH); U01CA062505 (NIH); U01CA069912 (NIH); U01CA070095 (NIH); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186689 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Glioma; Hematopoietic and Lymphoid Cell Neoplasm; Lymphoma; Metastatic Malignant Solid Neoplasm; Neuroendocrine Neoplasm; Recurrent Adult Soft Tissue Sarcoma; Recurrent Bladder Carcinoma; Recurrent Breast Carcinoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Colorectal Carcinoma; Recurrent Head and Neck Carcinoma; Recurrent Lung Carcinoma; Recurrent Malignant Solid Neoplasm; Recurrent Melanoma; Recurrent Pancreatic Carcinoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Prostate Carcinoma; Recurrent Renal Cell Carcinoma; Recurrent Thyroid Gland Carcinoma; Refractory Chronic Lymphocytic Leukemia; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage III Breast Cancer AJCC v7; Stage III Colorectal Cancer AJCC v7; Stage III Cutaneous Melanoma AJCC v7; Stage III Lung Cancer AJCC v7; Stage III Pancreatic Cancer AJCC v6 and v7; Stage III Prostate Cancer AJCC v7; Stage III Renal Cell Cancer AJCC v7; Stage III Soft Tissue Sarcoma AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Colorectal Cancer AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Lung Cancer AJCC v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Stage IV Prostate Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Glioma; Hematologic Neoplasms; Lymphoma; Neoplasm Metastasis; Neuroendocrine Tumors; Sarcoma; Urinary Bladder Neoplasms; Breast Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Colorectal Neoplasms; Lung Neoplasms; Melanoma; Pancreatic Neoplasms; Lymphoma, T-Cell, Cutaneous; Prostatic Neoplasms; Carcinoma, Renal Cell; Thyroid Neoplasms; Lymphoma, T-Cell | interventions — romidepsin; Depsipeptides; Lactones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (romidepsin) (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Pharmacological Study; Drug: Romidepsin

INTERVENTIONS:
Other: Pharmacological Study — Correlative studies
Drug: Romidepsin — Given IV
  Other Names: Antibiotic FR 901228; Depsipeptide; FK 228; FK-228; FK228; FR 901228; FR-901228; FR901228; Istodax; N-[(3S,4E)-3-Hydroxy-7-mercapto-1-oxo-4-heptenyl]-D-valyl-D-cysteinyl-(2Z)-2-amino-2-butenoyl-L-valine, (4->1) Lactone, Cyclic

SUMMARY:
This phase I trial studies the side effects and best dose of romidepsin in treating patients with lymphoma, chronic lymphocytic leukemia, or solid tumors with liver dysfunction. Romidepsin may stop the growth of cancer cells by entering the cancer cells and by blocking the activity of proteins that are important for the cancer's growth and survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety and tolerability of romidepsin given on days 1, 8, and 15 of a 28 day cycle to patients with varying degrees of liver dysfunction (mild, moderate and severe).

II. To establish the maximum tolerated dose (MTD) and appropriate dosing recommendations for romidepsin in such patients.

III. To characterize the pharmacokinetics (PK) of romidepsin in patients with varying degrees of liver dysfunction.

SECONDARY OBJECTIVES:

I. To explore correlations of the Child-Pugh classification of liver dysfunction with the observed toxicities and plasma PK of romidepsin administration.

II. To document any preliminary evidence of antitumor activity at tolerable doses of romidepsin in patients with varying degrees of liver dysfunction.

OUTLINE: This is a dose-escalation study.

Patients receive romidepsin intravenously (IV) over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed (at original diagnosis or subsequent recurrence or progression) lymphoma, chronic lymphocytic lymphoma (CLL) or solid tumor; patients with lymphoma or CLL must have radiologically or clinically evaluable disease, and be refractory to standard therapy as defined by relapse within 6 months of last treatment (see note below); patients with solid tumors must have radiologically or clinically evaluable disease that is metastatic, unresectable, progressive, or recurrent, and for which standard curative measures do not exist or are no longer effective

  * Patients with a liver mass, raised alpha-fetoprotein level (>= 500 ng/mL) and positive serology for hepatitis, consistent with a diagnosis of hepatocellular carcinoma will be eligible without the need for pathologic confirmation of the diagnosis
  * Patients with prostate cancer, renal cell cancer, neuroendocrine tumors, lung cancer, colorectal cancers, soft tissue sarcomas, glioma and thyroid cancer are excluded in the normal and mild cohorts due to a lack of efficacy in these tumor types in phase 2 studies; patients with breast, pancreatic, bladder, head and neck cancers, as well as melanoma and other malignancies are eligible
  * Note: patients with prostate cancer, renal cell cancer, lung cancer, colorectal cancers, soft tissue sarcomas, glioma and thyroid cancer are allowed to enroll in the moderate and severe cohorts provided the patients:

    * Sign a separate consent form which outlines the lack of efficacy observed in prior studies
    * Are consented to the study by a protocol-specified designee who is not their longitudinal oncologist; patients with neuroendocrine tumors are still excluded from the moderate and severe cohorts
  * Note: as romidepsin is approved for patients with relapsed or refractory peripheral T-cell lymphoma (PTCL) or cutaneous T cell lymphoma (CTCL), these patients would be eligible WITHOUT the requirement of having 'relapsed within 6 months of last treatment'
* Life expectancy of > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9 g/dL (transfusions and/or erythropoietin are permitted)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L (or platelet count >= 30 x 10^9 cells/L in patients with lymphoma or CLL if bone marrow disease involvement is documented)
* Creatinine =< twice upper limit institutional normal
* Patients with abnormal liver function will be eligible and will be grouped according to the criteria below

  * Group A (normal hepatic function)

    * Bilirubin =< upper limit of normal (ULN) and aspartate aminotransferase (AST) =< ULN
  * Group B (mild hepatic dysfunction)

    * B1: bilirubin =< ULN and AST > ULN
    * B2: bilirubin > ULN but =< 1.5 x ULN and any AST
  * Group C (moderate hepatic dysfunction)

    * Bilirubin > 1.5 x ULN to =< 3 x ULN and any AST
  * Group D (severe hepatic dysfunction)

    * Bilirubin > 3 x ULN and up to investigators discretion and any AST
  * Patients with active hemolysis should be excluded; no distinction will be made between liver dysfunction due to metastases and liver dysfunction due to other causes; registration laboratory investigations will be used to assign a patient to a hepatic function group; liver function tests should be repeated within 24 hours prior to starting initial therapy and may result in the patients' group assignment being altered if different to registration test results
* Patients with brain metastases who require corticosteroids or non-enzyme inducing anticonvulsants must be on a stable dose of corticosteroids and seizure free for 1 month prior to enrollment; patients with known brain metastases should have completed brain irradiation (whole brain or gamma knife) more than 4 weeks before starting the protocol; patients on enzyme inducing anticonvulsants are not eligible; note that patients should have had their steroids tapered to low dose (i.e. < 1.5 mg of dexamethasone/day) due to the potential for higher dexamethasone doses to induce CYP3A4
* Patients with biliary obstruction for which a stent has been placed are eligible, provided the shunt has been in place for at least 10 days prior to the first dose of romidepsin and the liver function has stabilized; two measurements at least 2 days apart that put the patient in the same hepatic dysfunction stratum will be accepted as evidence of stable hepatic function; there should be no evidence of biliary sepsis
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or PK of romidepsin will be determined following review of their case by the site principal investigator

  * Patients treated with any of the medications prohibited must discontinue their use at least 7 days prior to the first dose of romidepsin; certain other agents that interact with the CYP3A4 system may be used with caution
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; note: since romidepsin binds to the estrogen receptor, the effectiveness of estrogen containing contraceptives may be reduced
* Human immunodeficiency virus (HIV)-positive patients who are not receiving: agents with the potential for PK interactions with romidepsin or hepatotoxic antiretrovirals (nucleoside reverse-transcriptase inhibitors [NRTIs]: abacavir, didanosine, emtricitabine, lamivudine, stavudine, and zidovudine), dual protease inhibitor (PI)-based regimens except low-dose boosting with ritonavir, atazanavir, indinavir, maraviroc, and nevirapine may be eligible; additionally, the HIV-positive patients should have a cluster of differentiation (CD)4 count > 250/mm^3; if the specific cause of hepatic dysfunction is unknown, the patient should be worked up for other viral causes of hepatitis and their eligibility determined after consultation with the principal investigator
* Patients who have received prior romidepsin use are eligible
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had (prior to entering the study): major surgery and biologic/antibody therapies (including immunotherapies) are not permitted within 4 weeks of romidepsin administration; anti-cancer therapy including chemotherapy, radiotherapy, hormonal (with the exception of hormones for thyroid conditions), and other investigational agents will not be allowed within 14 days or five (5) half-lives (whichever is longer) prior to the first dose of romidepsin (6 weeks for nitrosoureas or mitomycin C); additionally, participants must have recovered to less than grade 2 clinically significant adverse effect(s)/toxicity(ies) of the previous therapy, with the exception of alopecia, unless approved by the principal investigator
* Patients with prostate cancer, renal cell cancer, neuroendocrine tumors, lung cancer, colorectal cancers, soft tissue sarcomas, glioma, and thyroid cancer are excluded in the normal and mild cohorts due to a lack of efficacy in these tumor types in phase 2 studies; patients with prostate cancer, renal cell cancer, lung cancer, colorectal cancers, soft tissue sarcomas, glioma and thyroid cancer are allowed to enroll in the moderate and severe cohorts only; patients with neuroendocrine tumors are still excluded from the moderate and severe cohorts
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to romidepsin, including cyclic tetrapeptide compounds
* Concurrent medications associated with a known risk of corrected QT interval (QTc) prolongation and/or Torsades de Pointes are not allowed within 2 weeks of initiation of study treatment; those medications listed as a possible risk for causing QTc prolongation and Torsades de Pointes will be allowed, although if an alternative medication can be substituted, that would be preferable; granisetron is an acceptable antiemetic on this study, but if a patient must take ondansetron, they may NOT take any other concomitant agents which might impact their QTc
* Thiazolidinedione agents such as rosiglitazone and pioglitazone are not permitted
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with current evidence of significant cardiovascular disease (New York Heart Association class III or IV cardiac disease), symptomatic congestive heart failure, dilated/hypertrophic or restrictive cardiomyopathy, myocardial infarction (within the past 6 months), unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medications for rate control for atrial fibrillation is allowed such as calcium channel blockers and beta-blockers, if stable medication for at least last month prior to initiation of romidepsin treatment and medication not listed as causing Torsades de Pointes), or evidence of acute ischemia on electrocardiogram (ECG); marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval > 450 msec*; long QT syndrome; the required use of concomitant medication that may cause Torsades de Pointes or may cause a significant prolongation of the QTc

  * Note: due to difficulties assessing QTc in patients with heart block, they may be eligible if deemed safe by a cardiologist; if a patient must take ondansetron as their antiemetic, their QTc may NOT be over 450 (no exception for patients with heart block)
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with this drug
* Warfarin is not permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of romidepsin in groups of patients with varying degree of hepatic dysfunction according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0 | 28 days
  Analyses will be descriptive in nature. The observed toxicities will be characterized by dose level within each category of liver dysfunction (mild, moderate, severe, and liver transplant). These results will be summarized in relation to what is known about romidepsin in a population without liver dysfunction (as defined in this protocol).
Dose-limiting toxicity of romidepsin in groups of patients with varying degree of hepatic dysfunction according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 5.0 | 28 days
  In order to define levels of hepatic impairment at which dose modifications of romidepsin are required, data will be combined across hepatic dysfunction groups to evaluate the association between toxicity, dose, and liver assay level(s). The outcome variable, drug tolerance and dose-limiting toxicities will be modeled as function of dose and liver assay using multivariate linear regression. Higher order terms of the predictor variables and interactions will be included if there is evidence of non-linear and/or non-additive associations.
Pharmacokinetic (PK) profile of romidepsin in patients with varying degrees of hepatic dysfunction using liquid chromatography-electrospray ionization tandem mass spectrometric method | 0, 1, 2, 3, 4, 4.25, 4.5, 5, 6, 8, 10, 24, and 48 hours after initiation of the infusion on day 1
  Pharmacokinetic variables will be tabulated and descriptive statistics calculated for each function group. Geometric means and coefficients of variation will be presented for maximum concentration and area under the curve for each group.

SECONDARY OUTCOMES:
Child-Pugh classification of hepatic dysfunction | Baseline
  Correlations of the Child-Pugh classification of hepatic dysfunction with the observed toxicities and plasma PK of romidepsin administration will be explored.
Antitumor activity assessed using Response Evaluation Criteria in Solid Tumors and the International Workshop Lymphoma Response Criteria | Up to 30 days
  Association of antitumor activity and romidepsin treatment will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Roisin M Connolly, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (12):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Case Western Reserve University, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada